CLINICAL TRIAL: NCT03011463
Title: Pharmacokinetic Interaction Between Trospium Chloride After Intravenous (2 mg) and Oral Administration (30 mg) With Ranitidine (300 mg p.o.) as an Inhibitor of OCT1 and With Clarithromycin (500 mg p.o.) as an Inhibitor of P-glycoprotein in 24 Healthy Subjects Genotyped for OCT1
Brief Title: Pharmacokinetic Interaction Between Trospium With an Inhibitor of OCT1 and of P-gp in Subjects Genotyped for OCT1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. R. Pfleger Chemische Fabrik GmbH (Industry)
Responsible Party: Principal Investigator, Tarek Roustom, top doctor, clinical trial center, University Medicine Greifswald
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: P334
Record Dates: First submitted 2017-01-02; First posted 2017-01-05 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Pharmacokinetics; Inhibition Enzyme; Drug Interaction Potentiation
MeSH Terms: interventions — trospium chloride; Ranitidine; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- trospium intravenous (Active Comparator): Intravenous infusion of 2 mg trospium chloride in 20 ml saline within 60 min and 240 ml tap water p.o.
  Interventions: Drug: intravenous infusion of 2 mg trospium chloride
- trospium oral (Active Comparator): Oral administration of 30 mg trospium chloride with 240 ml tap water
  Interventions: Drug: oral administration of 30 mg trospium chloride
- trospium intravenous with ranitidine (Active Comparator): Intravenous infusion of 2 mg trospium chloride in 20 ml saline within 60 min and oral administration of 300 mg ranitidine with 240 ml tap water
  Interventions: Drug: intravenous infusion of 2 mg trospium chloride; Drug: oral administration of 300 mg ranitidine
- trospium intravenous with clarithromycin (Active Comparator): Intravenous infusion of 2 mg trospium chloride in 20 ml saline within 60 min and oral administration of 500 mg clarithromycin with 240 ml tap water
  Interventions: Drug: intravenous infusion of 2 mg trospium chloride; Drug: oral administration of 500 mg clarithromycin
- trospium oral with ranitidine (Active Comparator): Oral administration of 30 mg trospium chloride together with 300 mg ranitidine with 240 ml tap water
  Interventions: Drug: oral administration of 30 mg trospium chloride; Drug: oral administration of 300 mg ranitidine
- trospium oral with clarithromycin (Active Comparator): Oral administration of 30 mg trospium chloride together with 500 mg clarithromycin with 240 ml tap water
  Interventions: Drug: oral administration of 30 mg trospium chloride; Drug: oral administration of 500 mg clarithromycin

INTERVENTIONS:
Drug: intravenous infusion of 2 mg trospium chloride — intravenous infusion of 2 mg trospium chloride in 20 ml saline within 60 min and 240 ml tap water p.o
  Arms: trospium intravenous; trospium intravenous with clarithromycin; trospium intravenous with ranitidine
Drug: oral administration of 30 mg trospium chloride — oral administration of 30 mg trospium chloride with 240 ml tap water
  Arms: trospium oral; trospium oral with clarithromycin; trospium oral with ranitidine
Drug: oral administration of 300 mg ranitidine — oral administration of 300 mg ranitidine with 240 ml tap water
  Arms: trospium intravenous with ranitidine; trospium oral with ranitidine
Drug: oral administration of 500 mg clarithromycin — oral administration of 500 mg clarithromycin with 240 ml tap water
  Arms: trospium intravenous with clarithromycin; trospium oral with clarithromycin

SUMMARY:
The purpose of the study is:

* to determine absolute bioavailability, input rates, distribution volume, renal and intestinal excretion of trospium in subjects with wild-type of SLC22A1 rs72552763 and rs12208357 and in subjects with homozygous variant alleles of SLC22A1 rs72552763 or rs12208357
* to determine absolute bioavailability, input rates, distribution volume and renal and intestinal excretion of trospium in subjects with wild-type alleles of SLC22A1 rs72552763 and rs12208357 after co-medication of 300 mg of the OCT1- inhibitor ranitidine
* to determine absolute bioavailability, input rates, distribution volume and renal and intestinal excretion of trospium in subjects with wild-type alleles of SLC22A1 rs72552763 and rs12208357 after co-medication of 500 mg of the P-glycoprotein- inhibitor clarithromycin
* to determine absolute bioavailability, input rates, distribution volume and renal and intestinal excretion of trospium in subjects with homozygous variant alleles of SLC22A1 rs72552763 or rs12208357 after co-medication of 500 mg of the P-glycoprotein- inhibitor clarithromycin.

ELIGIBILITY:
Inclusion Criteria:

* ethnic origin: Caucasian
* genotypes of OCT1: wild-type and homozygous variant alleles of SLC22A1 rs72552763 or rs12208357.
* body mass index: ≥ 18.5 kg/m² and ≤ 30 kg/m²
* good health as evidenced by the results of the clinical examination, ECG, and the laboratory check-up, which are judged by the clinical investigator not to differ in a clinical relevant way from the normal state (blood pressure between 110/70 and 140/90 for males and between 100/60 and 140/90 for females, heart rate over 50 bpm up to 90 bpm, laboratory values within the reference ranges as given actually by the laboratory and stored in the TMF)
* written informed consent

Exclusion Criteria:

* hepatic and renal diseases and/or pathological findings, which might interfere with pharmacokinetics and pharmacodynamics of the study medication (e.g. hepatic or renal dysfunction, obstruction of the urine flow with urinary retention by subvesical obstruction like benign prostatic hyperplasia, infections or tumors of the urinary tract)
* organic causes for polydipsia and pollakiuria
* existing cardiac or hematological diseases and/or pathological findings, which might interfere with the drug's safety, tolerability and/or pharmacokinetics (e.g. tachycardia, tachyarrhythmia, bradycardia, heart failure, coronary heart disease, disturbance of the stimulus conduction)
* pneumonia
* pharyngitis
* acute phorphyria
* hyperthyroidism
* galactose-intolerance, lactase deficiency or glucose-galactose malabsorption
* electrolyte disturbance
* gastrointestinal diseases and/or pathological findings (e.g. hiatus hernia with gastroesophageal reflux, stenosis, ulcera, severe chronic inflammatory bowel disease like ulcerative colitis or Crohn's disease, toxic megacolon), which might interfere with pharmacokinetics and pharmacodynamics of the study medication)
* autonomic neuropathy
* myasthenia gravis
* narrow-angle glaucoma
* drug or alcohol dependence
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day
* positive results in HIV, HBV and HCV screenings
* subjects who are on a diet which could affect the pharmacokinetics of the drugs (e. g. vegans, vegetarians)
* heavy tea or coffee drinkers (more than 1L per day)
* lactation, pregnancy test positive or not performed or women of child-bearing age without safe contraception as stated in the Note for Guidance on Non-clinical Safety Studies for the Conduct of Human Clinical Trials for Pharmaceutical (CPMP/ICH/286/95 modifications: implants, injectables, combined oral contraceptives, IUDs, sexual abstinence or vasectomised partner and barrier-methods only in combination with one of the aforementioned)
* subjects suspected or known not to follow instructions of the clinical investigators
* subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study
* subjects liable to orthostatic dysregulation, fainting, or blackouts
* participation in a clinical trial during the last 3 months prior to the start of the study
* less than 14 days after last acute disease
* less than 3 months after last blood donation
* any medication within 4 weeks prior to the intended first administration of the study medication which might influence functions of the gastrointestinal tract (e.g. laxatives, metoclopramide, loperamide, antacids, H2-receptor antagonists, proton pump inhibitors, anticholinergics)
* any other medication within two weeks prior to the first administration of the study medication, but at least 10-time the half-live of the respective drug (except oral contraceptives)
* intake of grapefruit or orange containing food or beverages within 14 days prior to administration of the study medication
* intake of poppy seed containing food or beverages within 14 days prior to administration of the study medication
* known allergic reactions to the active ingredients used, other H2-receptor antagonists, macrolide antibiotics or to constituents of the study medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
absolute bioavailability | up to 36 h after drug administration
  ratio oral over intravenous area under the concentration time curve normalized by given dose

SECONDARY OUTCOMES:
input rates | up to 36 h after drug administration
volume of distribution | up to 36 h after drug administration
renal excretion | up to 36 h after drug administration
intestinal excretion | up to 36 h after drug administration

IPD SHARING:
Plan to Share IPD: No